CLINICAL TRIAL: NCT03730363
Title: A Phase I Study of Pentamidine in Combination With Salvage Chemotherapy for Relapsed/Refractory Classical Hodgkin Lymphoma
Brief Title: Pentamidine + Salvage Chemo for Relapsed/Refractory Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reinhold Munker (Other)
Responsible Party: Sponsor-Investigator, Reinhold Munker, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18-HEM-13
Record Dates: First submitted 2018-10-26; First posted 2018-11-05 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
Keywords: Pentamidine; Salvage Chemotherapy
MeSH Terms: conditions — Hodgkin Disease | interventions — Pentamidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pentamidine + ICE (Experimental): Pentamidine, Ifosfamide, Carboplatin, and Etoposide (ICE) by IV Infusion.
  Interventions: Drug: Pentamidine

INTERVENTIONS:
Drug: Pentamidine — Pentamidine will be administered as an IV infusion on treatment day 1-3 of a 21-day cycle 3 cycles using 2, 3, and 4 mg/kg dose escalation schedules. Non-investigational agents will be administered as follows: Ifosfamide 5000 mg/m2, Carboplatin 5 area under curve (AUC), and Etoposide 100 mg/mg2.

SUMMARY:
Primary Objective:

To evaluate dose limiting toxicity and to determine the recommended phase 2 dose (RP2D) of pentamidine in combination with salvage chemotherapy with ifosfamide, carboplatin and etoposide (ICE) on a 3-weeks schedule in relapsed/refractory classical Hodgkin lymphoma (cHL).

Secondary Objective:

* To estimate the overall best treatment response at 5- and 16-weeks from study enrollment. Although the clinical benefit of these drugs in combination has not been established, offering this treatment may provide a therapeutic benefit. The patients will be carefully monitored for tumor response and symptom relief, in addition to safety and tolerability.
* To estimate the duration of response to the proposed combined therapy.
* To measure the protein of regenerating liver-3 (PRL-3) level of expression in patients at time of relapse.
* To measure circulating biomarkers of response (soluble CD30 (sCD30), and thymus and activation-related chemokine (TARC)) in serum samples collected throughout treatment and inhibition of (pSTAT, pAKT) in peripheral blood mononucleated cells (PBMC).

Exploratory Objective:

* To measure cell-free messenger RNA (cfmRNA) in peripheral blood.
* To measure cell-free DNA in peripheral blood

DETAILED DESCRIPTION:
The primary objective of this Phase I study is to determine the maximum tolerated dose (MTD) of Pentamidine. A two-stage continual reassessment method (CRM) will be employed to determine dose escalation levels and the maximum tolerated dose (MTD) of Pentamidine.

Specifically, a modified two-stage CRM will be employed with 2 patients per cohort at each dose level. The trial starts with an escalation design from the lowest dose (2 mg/kg) with a traditional 2+2 dose escalation method. After occurrence of the first DLT, dose assignment will be determined by the CRM (2 patients/per cohort) using empirical model with restrictions to avoid dose-skipping and escalation immediately after a toxicity outcome.

A maximum of 12 patients will be enrolled into the trial during the escalation phase. Once the MTD is reached, an additional 4 patients will be treated at this dose. Thus, 6 or more patients will be treated at the MTD.

The target DLT rate is 33% and the investigators choose to use 0.10, 0.20 and 0.33 as prior toxicity distribution. CRM simulations indicate optimal performance of this design with high dose recommendation probabilities (at least 48%) and more patients allocated to the correct dose

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Subjects with histologically confirmed relapse or refractory cHL who had received a front-line anthracycline-containing regimen.
* Subjects must have at least one measurable lesion >1.5cm as defined by the lymphoma response criteria.
* Subjects must have recovered from their last prior chemotherapy; if they have received an investigational agent, at least 5 half-lives must have expired to assure clearance of prior therapy.
* Prior radiation should have been completed at least 4 weeks prior to study Day 1.
* Toxicities related to prior therapy must have returned to Grade 1 or less except for alopecia. Peripheral neuropathy must be grade 2 or less.
* Adequate bone marrow function defined as: 1) Absolute neutrophil count ≥ 1000/µl and 2) Platelet count ≥ 50,000/µl
* Adequate organ function: 1) Creatinine Clearance (CrCl) >60 mL/min and 2) Aspartate Aminotransferase (AST) ≤ 3 upper limit normal (ULN), and Alanine Aminotransferase (ALT) ≤3 ULN, and Bilirubin ≤ 1.5 ULN (Unless they have Gillbert's disease)
* Ability to comply with the treatment, evaluations and required study follow-up.

Exclusion Criteria:

* Subjects with central nervous system involvement.
* Subjects with concomitant second malignancy (except adequately treated non-melanoma skin cancer, ductal carcinoma in-situ, superficial bladder cancer, prostate cancer or in situ cervical cancer) are excluded unless a complete remission was achieved at least 3 years prior to study entry and no additional therapy is required or anticipated.
* A serious uncontrolled medical disorder or active infection which impairs the ability of the subject to receive protocol therapy or whose control is jeopardized by the complication of this therapy.
* Prior organ allograft or allogeneic bone marrow transplantation.
* Positive for HIV (1/2) or known acquired immunodeficiency syndrome.
* Positive for hepatitis B Surface Ag, or antibody to hepatitis B core ag, or hepatitis C antibody or hepatitis C RNA in serum.
* Ejection fraction less than 45% in subjects with prior anthracycline therapy (measurement of ejection fraction is mandatory).
* Corrected QT interval (QTc) prolongation of more than 500.
* Women of reproductive age who are unwilling or unable to use an acceptable method to minimize the risk of pregnancy for the entire study period and for at least 18 weeks after the last dose of pentamidine.
* Women who are pregnant or breast-feeding.
* Women with a positive pregnancy test (serum assay) on enrollment or prior to pentamidine administration.
* Sexually active men not using birth control if their partners are women of reproductive age.
* Prisoner or subjects who are involuntarily incarcerated.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pentamidine and/or ifosfamide, carboplatin and etoposide.
* No investigational or commercial agents or therapies other than those specified by the protocol may be administered with the intent to treat the patient's malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 21 days
  Dose limiting toxicity (DLT) for hematological and non-hematological toxicities will be graded using National Cancer Institute (NCI) CTCAE Version 5.0

SECONDARY OUTCOMES:
Determine Efficacy: best overall response | Up to 112 days
  Individual best overall response at 5 and 16 weeks from enrollment, patients will be categorized as either a responder (complete response, partial response) versus nonresponders (stable disease, progressive disease).
Define the Duration of Response | Up to 112 days
  Duration of response as defined starting from the first occurrence of response until disease progression or death.
Identify Immunohistochemistry Biomarkers | Up to 112 days
  Immunohistochemistry staining of paraffin fixed tissue sample and peripheral blood will be done to assess the ability of pentamidine to inhibit its pharmacological target through PRL-3 expression.
Polymerase Chair Reaction (PCR) analysis of Biomarkers | Up to 112 days
  Digital PCR analysis of paraffin fixed tissue sample and peripheral blood will be done to assess PRL-3 expression and compare to the immunohistochemistry staining to determine the ideal testing modality for PRL-3 in cHL.
Identify Phosphorylation Biomarkers | Up to 112 days
  Pentamidine concentration/protein phosphorylation will be measured in PBMC and plasma samples collected throughout treatment.
Identify sCD30 and TARC Biomarkers | Up to 112 days
  Biomarkers: ELISA testing will be used to assess levels of sCD30 and TARC in serum samples collected prior to initiation of therapy and subsequent cycles.

OTHER OUTCOMES:
Measure cfmRNA Biomarkers | Up to 112 days
  Digital PCR analysis of the peripheral blood plasma will be used to measure cfmRNA during therapy
Measure Circulating-free DNA (cfDNA) Biomarkers | Up to 112 days
  digital PCR analysis of the peripheral blood plasma will be used to measure cfDNA during therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Hayder Saeed, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No